CLINICAL TRIAL: NCT03307915
Title: A Safety, Tolerability and Immunogenicity Study of 2 Different Regimens of Tetravalent Ad26.Mos4.HIV Prime Followed by Boost With MVA-Mosaic OR Ad26.Mos4.HIV Plus a Combination of Mosaic and Clade C gp140 Protein in HIV-1 Infected Adults on Suppressive ART
Brief Title: A Study of 2 Different Regimens of Tetravalent Ad26.Mos4.HIV Prime Followed by Boost With Modified Vaccinia Ankara (MVA)-Mosaic OR Ad26.Mos4.HIV Plus a Combination of Mosaic and Clade C gp140 Protein in Human Immunodeficiency Virus (HIV) Type 1 Infected Adults on Suppressive Antiretroviral Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); Ragon Institute of MGH, MIT and Harvard (Other); US Military HIV Research Program (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CR108372; VAC89220HTX1002 (Other: Janssen Vaccines & Prevention B.V.); IPCAVD-013 (Other: National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2017-09-25; First posted 2017-10-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Ad26.Mos4.HIV + MVA-Mosaic/Placebo (Experimental): Participants will receive adenovirus serotype 26-Mosaic 4 -Human Immunodeficiency Virus (Ad26.Mos4.HIV) 5*10^10 virus particles (vp) as intramuscular (IM) injection at Weeks 0 and 12 (1 injection) followed by modified Vaccinia Ankara-Mosaic (MVA-Mosaic) 10^8 Plaque-forming unit (pfu) and placebo as IM injection at Weeks 24 and 36 (2 injections).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: MVA-Mosaic; Drug: Placebo
- Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140 (Experimental): Participants will receive Ad26.Mos4.HIV, 5*10^10 vp as IM injection at Weeks 0 and 12 (1 injection) followed by both Ad26.Mos4.HIV 5*10^10 vp plus Clade C gp140 (125 microgram [mcg]) plus Mosaic gp140 (125 mcg) with aluminum phosphate adjuvant or an equivalent dose of a bivalent vaccine that includes both Clade C gp140 and Mosaic gp140, and aluminum phosphate adjuvant in a single vial, via IM injection at Weeks 24 and 36 (2 injections).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C gp140 + Mosaic gp140
- Group 3: Placebo (Placebo Comparator): Participants will receive 0.9 percent (%) saline as IM injection at Weeks 0, 12 (one injection) and at Week 24, 36 (two injections).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.Mos4.HIV — Participants will receive Ad26.Mos4.HIV 5*10^10 vp as 0.5 mL IM injection at Weeks 0, 12 in Group 1 and at Weeks 0, 12, 24, 36 in Group 2.
  Arms: Group 1: Ad26.Mos4.HIV + MVA-Mosaic/Placebo; Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Biological: MVA-Mosaic — Participants will receive MVA-Mosaic 10^8 pfu as IM injection at Weeks 24 and 36.
  Arms: Group 1: Ad26.Mos4.HIV + MVA-Mosaic/Placebo
Biological: Clade C gp140 + Mosaic gp140 — Participants will receive both Clade C gp140 125 mcg plus Mosaic gp140 125 mcg (250 mcg coformulated with Aluminum phosphate adjuvant) OR an equivalent dose of a bivalent vaccine that includes both Clade C gp140 and Mosaic gp140, and aluminum phosphate adjuvant in a single vial, via IM injection at Weeks 24 and 36.
  Arms: Group 2: Ad26.Mos4.HIV + Clade C gp140 + Mosaic gp140
Drug: Placebo — Participants will receive matching placebo as IM injection at Weeks 24, 36 in Group 1 and at Weeks 0, 12, 24, 36 in Group 3.
  Arms: Group 1: Ad26.Mos4.HIV + MVA-Mosaic/Placebo; Group 3: Placebo

SUMMARY:
The primary purpose of this study is to assess safety/tolerability of 2 different prime/boost regimens containing adenovirus serotype 26 (Ad26).Mos4.HIV, Modified Vaccinia Ankara (MVA) -Mosaic or adjuvanted Mosaic and Clade C gp140 in Human immunodeficiency virus type 1 (HIV-1)-infected participants on suppressive antiretroviral treatment (ART).

ELIGIBILITY:
Inclusion Criteria:

* Each participant must have documented Human immunodeficiency virus type1 (HIV-1) infection
* Each participant must be on suppressive antiretroviral treatment (ART) for at least 48 weeks prior to randomization and on stable suppressive ART for at least 4 weeks prior to screening. Changes in antiretrovirals (ARVs) can be made for safety/tolerability reasons only until 4 weeks prior to screening
* Each participant must have started ART outside of the acute or early phase of infection
* Each participant must have a plasma HIV ribonucleic acid (RNA) less than (<) 50 copies/ milliliter (mL) at screening and at least one documented evidence of plasma HIV RNA <50 copies/mL after the last ART change. In case of ART change within the 48 weeks prior randomization, at least one additional more recent documented plasma HIV RNA <50 copies/mL is required. One blip of HIV RNA greater than (>)50 and <200 copies/mL within 24 weeks prior to screening is acceptable, provided that the 2 most recent (after last ART change, tested before and/or during screening) HIV RNA results are <50 copies/mL
* Each participant must be medically stable as confirmed by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening

Exclusion Criteria:

* Anyone who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study, or within 3 months after the last vaccination
* Anyone with contraindication to intramuscular injections and blood draws example, bleeding disorders
* Anyone with acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0ºC (degree centigrade) within 24 hours prior to the first dose of study vaccine; enrollment at a later date is permitted
* Anyone with a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Anyone with a history of an underlying clinically significant acute or uncontrolled chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Anyone with a history of Acquired Immunodeficiency Syndrome (AIDS)-defining illness according to Centers for Disease Control and prevention (CDC) criteria based on available medical history and assessed by the investigator as clinically relevant. A case summary for every participant with AIDS-defining illnesses assessed by the investigator as clinically irrelevant must be provided to the sponsor and Protocol Safety Review Team (PSRT), who will determine eligibility on a case-by-case basis prior to randomization
* Anyone with a history of CD4+ less than (<) 200 cells per millimeter cube (cells/mm^3), based on available medical history and assessed by the investigator as clinically relevant. A case summary for every participant with history of CD4+ <200 cells/mm^3 assessed by the investigator as clinically irrelevant must be provided to the sponsor and PSRT, who will determine eligibility on a case-by-case basis prior to randomization
* Anyone with chronic active hepatitis B (measured by hepatitis B surface antigen test) or active hepatitis C (measured by hepatitis C virus [HCV] antibody test; if positive, HCV RNA polymerase chain reaction test will be used to confirm active versus past HCV infection) or syphilis infection that has not been effectively treated. Positive syphilis serology due to past effectively treated infection is not exclusionary
* Anyone who received or plans to receive: a) licensed live attenuated vaccines within 28 days before or after planned administration of any of the study vaccinations; b) other licensed (not live) vaccines - within 14 days before or after planned administration of any of the study vaccinations
* Anyone who received an investigational drug or used an invasive investigational medical device within 30 days or received an investigational vaccine within 6 months before the planned administration of the first dose of study vaccine. Receipt of prophylactic or therapeutic HIV vaccine candidate at any time is always exclusionary. Exceptions: Participants can be included where the vaccine received was subsequently licensed. Participants with proof of having received only a placebo vaccine can also be included

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local Adverse Events (AEs) as a Measure of Safety and Tolerability | 7 days post-vaccination (approximately up to 37 weeks)
  Solicited local AEs: erythema, swelling/induration, and pain/tenderness will be assessed.
Percentage of Participants With Solicited Systemic AEs as a Measure of Safety and Tolerability | 7 days post-vaccination (approximately up to 37 weeks)
  Solicited systemic AEs: fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills will be assessed.
Percentage of Participants With AEs as a Measure of Safety and Tolerability | Approximately up to 96 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Total IgG and Subclass Specific Antibody Titer | Up to post-vaccination follow-up period until Week 96
  Total immunoglobulin G (IgG) and subclass (IgG1-4) specific antibody titers (binding antibody) to envelope (Env) proteins representing Clades A, B, and C, as well as Mosaic antigens.
Antibody Functionality Assessment by Antibody-dependent Cell-mediated Phagocytosis (ADCP) | Up to post-vaccination follow-up period until Week 96
  Antibody functionality assessment will be assessed by antibody-dependent cell-mediated phagocytosis (ADCP) assay.
Magnitude of T-cell Responses as Measured by Intracellular Cytokine Staining (ICS) Assay | Up to post-vaccination follow-up period until Week 96
  Intracellular cytokine staining (ICS) assays with Env, group-specific antigen (Gag), and/or polymerase (Pol)-peptide pools will be used to determine the magnitude of T-cell responses elicited.
Functionality of T-cell Responses as Measured by ICS Assay | Up to post-vaccination follow-up period until Week 96
  ICS assays with Env, Gag, and/or Pol-peptide pools will be used to determine the functionality of T-cell responses elicited.
Phenotype of T-cell Responses as Measured by ICS Assay | Up to post-vaccination follow-up period until Week 96
  ICS assays with Env, Gag, and/or Pol-peptide pools will be used to determine the phenotype of T-cell responses elicited.
Frequency of Epitope Recognition by Enzyme-Linked Immunospot (ELISPOT) | Up to post-vaccination follow-up period until Week 96
  Assays of peptide pool sets covering the Gag, Env or Pol will be evaluated by standard enzyme linked immunospot assay (ELISPOT).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States